CLINICAL TRIAL: NCT04210479
Title: Bladder Filling in Cesarean Hysterectomy for Placenta Percreta: A Randomized Trial
Brief Title: Comparison of Bladder Filling vs. Non-Filling in Cesarean Hysterectomy for Placenta Percreta
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hatem AbuHashim (Other)
Responsible Party: Sponsor-Investigator, Hatem AbuHashim, Professor, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MS.19.12.939
Record Dates: First submitted 2019-12-21; First posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Filled-bladder (Experimental): Bladder filling with 300ml diluted methylene blue.
  Interventions: Procedure: Filled-bladder
- non filled-bladder (Active Comparator)
  Interventions: Procedure: non filled-bladder

INTERVENTIONS:
Procedure: Filled-bladder — Urinary bladder filling with 300 ml diluted methylene blue
  Arms: Filled-bladder
Procedure: non filled-bladder — Pull up the empty (non-filled) urinary bladder using Allis forceps
  Arms: non filled-bladder

SUMMARY:
The placenta accreta spectrum (PAS) which includes accreta, increta, and percreta represents a significant obstetric challenge. PAS complicates as many as 1 per 500 pregnancies and this risk is increased with prior cesarean deliveries. Antenatal diagnosis of PAS allows for multidisciplinary planning and delivery before the onset of labor and/or vaginal bleeding. This approach has reduced maternal morbidity rates. including less blood loss, fewer transfusion requirements and, intraoperative urinary tract injury as well as improve fetal outcome.

Ultrasound evaluation is the recommended first-line modality for diagnosing PAS. Ultrasound features suggestive of PAS include loss of the normal retroplacental clear zone, attenuation of the uterine-bladder interface, reduced retroplacental myometrial thickness, presence of intraplacental lacunar spaces, and bridging vessels between the placenta and bladder. A systematic review reported that the antenatal diagnosis of PAS significantly lowered the rate of urinary tract injury (from 63% to 39%) during cesarean hysterectomies in these cases.

Unlike other elective cesarean hysterectomies, cesarean hysterectomy with a placenta previa increta/percreta, is more difficult. There is a greater need to both keep a margin from the vascular cervical-placental mass and simultaneously protect the urinary bladder. Case series reported that bladder filling helps the surgeon to more clearly identify the planes of dissection and secure the engorged aberrant vessels, thereby reduces bladder injury. Accordingly, a prospective randomized study in pregnant patients with placenta previa increta/percreta undergoing elective cesarean hysterectomy will be conducted to address this important issue.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in their third trimester (35-37 W).
* Placenta previa accreta spectrum identified by the Ultrasound (low lying anterior or major degree anterior).
* With at least one prior cesarean section.
* Elective cesarean hysterectomy.
* Evidence of gross placental invasion at the time of surgery (FIGO grade 3a.

Exclusion Criteria:

* Patients undergoing conservative treatment.
* Emergency cesarean hysterectomy.
* No evidence of gross placental invasion at the time of surgery.
* Posterior placenta.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-01-15 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of urinary bladder injury | Intra-operative (i.e. during surgery).
  Unintentional bladder injury during elective cesarean hysterectomy

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Abu Hashim, MD. FRCOG. PhD, Study Chair — Faculty of Medicine, Mansoura University; Mostafa Aboelenin, MBBCh, Principal Investigator — Samnoud General Hospital

REFERENCES:
- [Result] Matsubara S. Caesarean hysterectomy for placenta praevia accreta: filling the bladder technique to identify an appropriate bladder separation site. J Obstet Gynaecol. 2013 Feb;33(2):163-4. doi: 10.3109/01443615.2012.740525. No abstract available. PMID 23445140